CLINICAL TRIAL: NCT06918496
Title: A Prospective ClinicaL investigatiOn Evaluating Prophylactic Sealing of sUture Lines Using the NE'X Glue R-eco Surgical AdhesivE in Cardiac and (Cardio)Vascular Anastomotic Repair Procedures
Brief Title: Prophylactic Suture Line Sealing With NE'X Glue R-eco in Cardiac and Vascular Surgery
Acronym: CLOSURE
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Grena Biomed Limited (Industry)
Collaborators: Archer Research (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: CIV-24-12-050294
Record Dates: First submitted 2025-03-21; First posted 2025-04-09 (Actual); Last update posted 2025-04-09 (Actual); Status verified 2025-04

CONDITIONS: Aortic Aneurysm; Aortic Aneurysm Abdominal; Valve Stenoses, Aortic; Valve Regurgitation, Mitral; Valve Regurgitation, Tricuspid; Aneurysm of Ascending Aorta; Aneurysm Abdominal; Artery Diseases, Peripheral; Ventricular Aneurysm; Coronary Artery Disease; Valve Aortic Regurgitation; Aortic Aneurysms Arch; Aortic Aneurysms Descending; Aortic Aneurysms Thoracoabdominal
Keywords: prophylactic sealing of suture lines; Surgical glue; cardiac and (cardio)vascular anastomotic repair procedures; grafts; NE'X Glue R-eco surgical adhesive
MeSH Terms: conditions — Aortic Aneurysm; Aortic Aneurysm, Abdominal; Aortic Valve Stenosis; Mitral Valve Insufficiency; Tricuspid Valve Insufficiency; Aneurysm, Ascending Aorta; Peripheral Arterial Disease; Coronary Artery Disease; Aortic Valve Insufficiency; Aneurysm, Aortic Arch; Aortic Aneurysm, Thoracoabdominal | interventions — Transdermal Patch

STUDY DESIGN:
Intervention Model Description: Pre-market, pivotal, commercial, prospective, single-arm, interventional, multicenter clinical investigation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Single-arm (Experimental): A single-arm design is selected, providing data about safety and clinical effectiveness of the NE'X Glue R-eco of which are to be compared to established data available in the literature
  Interventions: Device: Surgical placement of a prosthetic or biologic graft (patch), or an allograft for cardiac and (cardio)vascular repair.

INTERVENTIONS:
Device: Surgical placement of a prosthetic or biologic graft (patch), or an allograft for cardiac and (cardio)vascular repair. — Suture line bleeding in cardiac and vascular reconstruction poses significant risks, including morbidity, mortality, and complications related to blood loss and transfusion. Advances in surgical techniques have improved hemostasis but may not suffice, especially in patients on anticoagulant or antiplatelet medications or those using synthetic graft materials.
  Surgical adhesives are valuable adjuncts to standard hemostatic techniques, aiming to prevent postoperative bleeding and its associated complications. NE'X Glue R-eco, a novel surgical adhesive, utilizes recombinant human serum albumin (rHSA) and glutaraldehyde (GA) for suture line sealing. It is similar to BioGlue®, which uses bovine serum albumin (BSA) and GA, and has proven safety and benefits.
  Distinguishing Features of NE'X Glue R-eco:
  Composition: Uses rHSA expressed in plants, offering improved biocompatibility and reduced risk of allergic reactions.
  Bonding Strength: Demonstrates high bonding strength in tests, comparab

SUMMARY:
This clinical study aims to evaluate the effectiveness and safety of using NE'X Glue R-eco to seal suture lines. The adhesive will be applied to reduce the risk of suture line bleeding in cardiac or vascular repair surgeries, a prosthetic or biologic graft, patch, or allograft.

The effectiveness of the adhesive will be assessed after restoring blood flow.

DETAILED DESCRIPTION:
Suture line bleeding is a common issue in cardiovascular surgeries, leading to serious complications and increased costs. Effective management is crucial to prevent morbidity, fatal consequences, and the need for reoperation, which has high mortality rates. Blood transfusions carry risks, and patients who avoid them tend to recover better. Advances in surgical techniques and the use of anticoagulants have increased the need for robust methods to prevent suture line bleeding.

Surgical adhesives are becoming standard practice to prevent air and liquid leaks during surgeries. Different classes of adhesives, such as cyanoacrylates, polyethylene glycol polymers, bovine serum albumin (BSA) and glutaraldehyde mixtures, gelatin and thrombin sealants, and fibrin sealants, offer various advantages and disadvantages.

Most cyanoacrylate sealants are used externally due to risks of infection, cytotoxicity, and tissue necrosis when used internally. They are effective for closing skin incisions, trauma wounds, and providing a microbial barrier over closed wounds. Polyethylene glycol hydrogel adhesives are valued for their biocompatibility, degradability, and tunable mechanical properties, acting as both fluid barriers and hemostatic agents. However, they can cause significant post-polymerization swelling. Fibrin sealants, derived from blood, are used as hemostatic agents in cardiac, liver, and splenic surgeries. They carry risks of transmitting infections and air or gas embolism. Gelatin and thrombin mixtures are versatile hemostatic agents used in various surgeries, including delicate structures like nerves, due to their low toxicity.

The last class of surgical adhesives includes mixtures of bovine serum albumin (BSA) and glutaraldehyde (GA) or polyaldehyde. In BioGlue® (CryoLife Inc.) and PREVELEAKTM (Baxter Advanced Surgery), BSA crosslinks with extracellular proteins to form a mechanical seal independent of the coagulation system. NE'X Glue R-eco, a new adhesive by Grena BioMed Limited, is similar to BioGlue® but uses recombinant human serum albumin (rHSA) instead of BSA. Both adhesives use a double-chambered syringe for controlled application.

BioGlue® has proven biocompatibility, reliability, and safety, with minor differences in external shape compared to NE'X Glue R-eco. BioGlue® has passed extensive biological evaluations and animal studies, demonstrating its effectiveness in surgical repairs.

Analytical and functional tests have shown that NE'X Glue R-eco has adequate bonding strength and similar chemical properties to BioGlue®. The safety and benefits of these adhesives have been demonstrated in various studies. This pivotal study aims to evaluate the efficacy and safety of NE'X Glue R-eco for sealing suture lines. The study will assess immediate and delayed suture line sealing, sealing time, use of additional agents, product handling, blood loss, use of blood replacement products, anticoagulant/antiplatelet medication intake, device deficiencies, and peri- and postoperative complications and re-interventions.

The primary objective of this study is to evaluate the immediate sealing of suture lines using NE'X Glue R-eco. The secondary objective is to assess the overall efficacy and safety of NE'X Glue R-eco for prophylactic suture line sealing.

This clinical investigation uses a single-arm, non-randomized design to evaluate the safety and effectiveness of surgical adhesives in cardiac and vascular procedures. Strict inclusion and exclusion criteria prevent bias, ensuring participants represent the general population needing these surgeries. Exclusion criteria include hypersensitivity, active infection, vasculitis, bleeding disorders, immune suppression, and refusal of blood transfusions. Clinical Research Associates will monitor the study and report any deviations.

Participants will be followed for up to 3 months post-surgery to document potential complications such as inflammatory responses, allergic reactions, tissue necrosis, vessel obstruction, thrombosis, and more. This follow-up period allows for clear documentation of safety and effectiveness.

Patients undergoing large vessel and cardiac repair, arterial reconstruction, or arteriovenous graft formation with prosthetic or biologic grafts (patches) or allografts will be included in this study. Data will be collected from 60 patients at sites in Belgium and Poland. Inclusion and exclusion criteria ensure a diverse participant cohort reflective of the broader population. Minors, pregnant women, and breastfeeding women are excluded. Female participants of childbearing age must use contraception and undergo pregnancy testing. Incapacitated patients may be included if their medical condition prevents informed consent. Follow-up monitoring will be conducted for up to 3 months post-procedure.

ELIGIBILITY:
Inclusion Criteria:

* Patient ≥ 18 years of age at study entry.
* Patient is scheduled for open procedures for surgical placement of a prosthetic or biologic graft (patch) or an allograft for cardiac and (cardio)vascular anastomosis repair. Emergency, transplantation and minimally invasive procedures are excluded. Patients receiving long-term anticoagulation, including antiplatelet agent, are included. Choice of graft is at the discretion of the surgeon.
* Patient is willing and able to be contacted for up to 3 months (± 14 days) follow-up.
* Patient or legal representative and investigator signed and dated the informed consent form prior to the index-procedure.

Exclusion Criteria:

* Patient has a known hypersensitivity, contraindication, or allergic reaction to albumin or glutaraldehyde.
* Patient has a history of bleeding diathesis or coagulopathy.
* Presence of active infection or contamination in the to be grafted area or the vicinity.
* Known vasculitis in the to be grafted area.
* Patient takes immune suppressive medication like prednisone resulting in weakening of the vessel wall.
* Patient is refusing blood transfusion.
* Patient or legal representative is unable / unwilling to provide informed consent.
* Patient is unable to comply with the protocol or proposed follow-up visits.
* Female patient is pregnant, lactating, or planning pregnancy during the clinical investigation.
* Female participants of childbearing age must agree to use safe contraception (e.g., intrauterine devices, hormonal contraceptives: contraceptive pills, implants, transdermal patches hormonal vaginal devices, injections with prolonged release, abstinence).
* Patients who are currently enrolled in another clinical study, or have recently participated in a clinical study, that could potentially interfere with the outcomes or introduce bias into the results of the current study (as determined by the investigator). This includes studies involving investigational drugs, medical devices, or other interventions that could impact the safety, efficacy, or scientific integrity of this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-30 (Estimated); Primary Completion 2026-03-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Evaluate immediate suture line sealing using NE'X Glue R-eco. | From index-procedure until end of participation in the study at 3 months
  Proportion of patients/anastomoses with immediate suture line sealing by NE'X Glue R-eco, evidenced by lack of clinically significant bleeding (bleeding status is 'No bleeding' or 'Oozing'), as judged by the surgeon immediately after clamp release.
  Clamp release is performed 2 minutes after the application of the adhesive. Bleeding is classified into one of four categories: 1. No bleeding, 2. Oozing, 3. Fast flow, 4. Spurting, where 1 and 2 will be considered as 'no clinically significant bleeding' and 3 and 4 as 'bleeding'.
  Sealing time refers to the time the anastomotic site is completely sealed, that is, the last time point in which bleeding status equaled 'No bleeding' and 'Oozing'.
  Immediate sealing means the sealing time is 0. For patients with multiple anastomoses, immediate suture line sealing should occur in all for the patient to have no clinically significant bleeding at sealing time 0.

SECONDARY OUTCOMES:
To determine the proportion of patients/anastomoses with suture line sealing using NE'X Glue R-eco, measured at 1, 3, 5, and 10 minutes after clamp release (timed with a calibrated stop watch). | During the index-procedure
  The cases where the investigator choses to intervene and use additional methods to achieve hemostasis will be defined as 'bleeding'. For patients with more than one anastomotic site treated, the site with the longest time to hemostasis was used for these analyses. If fast flow or spurting, the surgeon may use additional agents for hemostasis before the 10 minutes are up to guarantee the safety of the patient.
To determine the elapsed time from clamp release to hemostasis (sealing time) recorded per site. | During the index-procedure
  Sealing time refers to the time the anastomotic site is completely sealed, that is, the last time point in which bleeding status equaled 'No bleeding' and 'Oozing'.
  Anastomoses where the investigator choses to intervene and use additional methods to achieve hemostasis will not be included in this analysis. Any time to hemostasis that was >10 minutes was treated as 10 minutes in the analysis.
To determine the use of any additional methods to achieve hemostasis (including pledgets, sutures, hemostatic devices, antifibrinolytic agents, thrombin glues, fibrin glues, etc.) (type and quantity). | During the index-procedure
  For patients with more than one anastomotic site treated, each patient will be classified as having had an additional agent or not.
To determine the product handling and performance of NE'X Glue R-eco | During the index-procedure
  By documenting the following outcomes, using the following four possible responses: excellent, good, fair or poor.
  * Ease of preparing
  * Performance of the delivery system
  * Gel rate
  * Adhesiveness
To determine device deficiencies | During the index-procedure
  These device deficiencies may include, but are not limited to
  * Failure of adhesive to adhere to tissue
  * Failure of sealing
  * Device malfunction
To determine blood loss during the first 24-48 hours post-surgery | During the first 24-48 hours post-surgery (post index-procedure)
  Estimated blood loss by visual inspection or gravimetric method.
To determine the intake of anticoagulant/antiplatelet medication | From screening until end of participation in the study at 3 months
  The intake will be documented at screening, index-procedure, discharge, 5 weeks follow-up and 3 months follow-up.
To determine the intra-operative and post-operative complication rate | From index-procedure until end of participation in the study at 3 months
  Complications may include, but are not limited to:
  * Hypersensitivity reaction such as swelling or edema at the application site
  * Application of adhesive to tissue not targeted for procedure resulting in a complication
  * Local tissue necrosis
  * Mineralization of tissue
  * Infection
  * Thrombosis and thromboembolism
  * Intra- and post-operative significant bleeding, defined as a steady stream of blood that would not resolve without intervention
  * Ischemia
  * Myocardial infarction
  * Neurological deficit
  * Organ system failure
  * Paraplegia
  * Renal dysfunction/failure
  * Respiratory dysfunction/failure
  * Stroke or cerebral infarction
  * Other complications related to cardiac and (cardio)vascular procedures
Return to the operating room (re-interventions) within 3 months. | From index-procedure until end of participation in the study at 3 months
Mortality / Decease | From index-procedure until end of participation in the study at 3 months
To determine the use of any blood replacement products | From index-procedure until end of participation in the study at 3 months
  Type and quantity will be documented

CONTACTS AND LOCATIONS:
Locations (2):
- Jessa Hospital, Hasselt, Limburg, Belgium
- Klinika Kardiochirurgii i Transplantologii, Warsaw, Poland